CLINICAL TRIAL: NCT05315336
Title: L-DEP/DEP Regimen and PD-1 Antibody as a Treatment for Relapse/Refractory EBV Associated Hemophagocytic Lymphohistiocytosis (HLH)
Brief Title: L-DEP/DEP Regimen and PD-1 Antibody as a Treatment for Relapse/Refractory EBV-HLH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Department of Hematology, Beijing Friendship Hospital, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-DEP, PD-1, HLH
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Hemophagocytic Lymphohistiocytosis; DEP; L-Asparaginasum; PD-1 antibody
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Intervention Model Description: All patients with R/R EBV- HLH receive DEP combine with PD-1 antibody as an treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-DEP and PD-1 antibody (Experimental): Doxorubicin (doxorubicin hydrochloride liposome injection) 25 mg/m2 day 1; etoposide 100 mg/m2 was administered day1; methylprednisolone 2mg/kg days 1 to 3,then 0.25mg/kg day 4 to 14; PD-1 antibody injection 200mg day 5; L-asparaginases 6000iu/m2 day2, day4. This regimen was repeated after 2 weeks.
  Interventions: Drug: L-DEP and PD-1 antibody

INTERVENTIONS:
Drug: L-DEP and PD-1 antibody — Doxorubicin (doxorubicin hydrochloride liposome injection) 25 mg/m2 day 1; etoposide 100 mg/m2 was administered day1; methylprednisolone 2mg/kg days 1 to 3,then 0.25mg/kg day 4 to 14; PD-1 antibody injection 200mg day 5; L-asparaginases 6000iu/m2 day2, day4. This regimen was repeated after 2 weeks.

SUMMARY:
This study aimed to investigate the efficacy and safety of L-DEP (L-Asparaginasum, liposomal doxorubicin, etoposide and methylprednisolone) together with PD-1 antibody as an treatment for relapse/refractory EBV associated hemophagocytic lymphohistiocytosis.

DETAILED DESCRIPTION:
PD-1 antibody added to the DEP regimen （with or without asparaginases） in EBV-HLH

ELIGIBILITY:
Inclusion Criteria:

1. Meet hemophagocytic lymphohistiocytosis (HLH)-04 diagnostic criteria;patients were diagnosed with EBV associated HLH (EBV-HLH).
2. EBV-DNA in peripheral blood or EBER in tissue were positive.
3. Treated with HLH-94 no less than 2 weeks before enrollment and did not achieve at least partial response
4. The patient is expected to be unable to undergo allogeneic hematopoietic stem cell transplantation in the short term due to various reasons (physical status, economic reasons, donor reasons, etc.)
5. The expected survival time is more than 1 month.
6. Age ≤ years old, gender is not limited.
7. Serum creatinine ≤ 1.5 times normal；After infusion, fibrinogen can be corrected to ≥0.6g/L.
8. Serum human immunodeficiency virus(HIV) antigen or antibody negative； Hepatitis C virus (HCV) antibody is negative, or HCV antibody is positive, but HCV RNA is negative；HBV copies less than 1E+03 copies/ml.
9. The left ventricular ejection fraction (LVEF) was normal.
10. No uncontrollable infection.
11. Contraception for both male or female.
12. Informed consent obtained.

Exclusion Criteria:

1. Allergic to doxorubicin and/or etoposide and/or PD-1 antibody Injection
2. Severe myocardial injury, myocardial enzymes CK, CK-MB increased more than 3 times ULN (upper limit of normal)
3. Heart function above grade II (NYHA).
4. Thyroid dysfunction
5. Serious mental illness;
6. Active hemorrhage of internal organs
7. Previously received L-DEP regimen for HLH-targeted treatment, but the treatment was ineffective or relapsed
8. Accumulated dose of doxorubicin above 300mg/m2 or epirubicin above 450mg/m2
9. Participate in other clinical research at the same time.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment response | Change from before and 2,4,6 and 8 weeks after initiating DEP combine with PD-1 antibody therapy
  The primary observed endpoint is the objective remission rate (ORR): cases that include complete remission (CR) and partial remission (PR).CR was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT). PR was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.

SECONDARY OUTCOMES:
EBV-DNA | Change from before and 2,4,6 and 8 weeks after initiating DEP combine with PD-1 antibody therapy
  Outcome of patients with EBV-HLH
Survival | 3 months after the intervention
  Outcome of patients with EBV-HLH
Adverse events that are related to treatment | 2,4,6 and 8 weeks after initiating DEP combine with PD-1 antibody therapy
  Incidence of events that are related to treatment including myelosuppression, infection, bleeding and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China